CLINICAL TRIAL: NCT01474018
Title: QR-Bromocriptine as an Adjunct to Insulin and Metformin in the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QR-Bromo
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin + Insulin (No Intervention): 5 patients to continue on usual type 2 diabetic treatment consisting of 70/30 insulin, metformin and exercise and nutrition counseling.
- QR-Bromocriptine +metformin+insulin (Experimental): study drug add-on the usual therapy
  Interventions: Drug: QR-bromocriptine

INTERVENTIONS:
Drug: QR-bromocriptine — The study drug is added-on to patients on existing type 2 diabetes treatment with insulin +metformin+exercise/nutritional counseling. The study drug is titrated up starting at one 0.8mg tab daily for 1 week, then 2 (0.8mg) tablets for week 2, then 3 tablets for week 3, then 4 tablets for week 4, then 5 tablets for week 5, then six tablets for week 6 (total 4.8). The limiting factor is nausea at which point the patients will back down the highest tolerated dose and continue on that dose for the remainder of the 6 months of the study.
  Other Names: NDC 6801225820; Cycloset (brand)
  Arms: QR-Bromocriptine +metformin+insulin

SUMMARY:
QR-Bromocriptine as an add-on treatment to insulin and metformin in the management of type 2 diabetes will result in improved glycemic control, reduced exogenous insulin requirement, increased lean fat mass and improved pancreatic beta-cell function.

DETAILED DESCRIPTION:
To assess improvement in glycemic control, reliance on exogenous insulin, improvements in lean body mass composition, and improvements in pancreatic beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, age 30 to 65 years of age,
2. Clinical diagnosis of type 2 diabetes at least 6 months prior to enrollment,
3. Stable on current treatment consisting of either human or recombinant multi-dose insulin therapy (MDI) with metformin,
4. HbA1c of 7.5-12%, inclusive,
5. Demonstrated willingness to check and record blood glucose readings at seven time points as instructed in the study protocol.
6. Medically controlled hypertension, at least on one anti-hypertensive
7. Medically controlled hyperlipidemia, on or off cholesterol-lowering therapy
8. BMI >30

Exclusion Criteria:

1. Pregnancy or Lactating,
2. Type 1 Diabetes,
3. Concomitant use of forbidden medications: prescription sympathomimetics (within seven days of screening), ergot alkaloid derivatives, and anti-migraine medications,
4. Patients with history of drug or alcohol abuse within 3 years of enrollment,
5. Patients at risk for hypotension, including those who have:

   * Recent blood donation within 30 days of enrollment,
   * A history of syncopal migraines, or
   * Significant gastroparesis or orthostatic hypotension which could signify advanced autonomic neuropathy.
6. Uncontrolled mental illness especially with history of psychosis,
7. Any severe, uncontrolled or terminal medical condition which the investigator feels would interfere with the patient's ability to participate and comply with the study protocol,
8. Serum creatinine >1.4mg/dL in females or >1.5mg/dL in males that would preclude the patient from taking metformin,
9. LFTs elevated >3x upper limit of normal,
10. Patients working rotating, varying or night shifts, or
11. Patient with circumstances or abnormalities (e.g. blindness or history of non-compliance) that would interfere with the interpretation of safety or efficacy data or completion of the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Raskin, MD, Principal Investigator — UTexas Southwestern
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin + Insulin: 5 patients to continue on usual type 2 diabetic treatment consisting of 70/30 insulin, metformin and exercise and nutrition counseling.
  Study has completed
Period: Overall Study
Arm/Group | Metformin + Insulin | QR-Bromocriptine +Metformin+Insulin
Started | 5 | 10
Completed | 5 (Writing paper) | 7
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients age 30-65 years with the clinical diagnosis of T2DM on multiple daily injections of insulin plus metformin and HbA1c between 7.5-12.0% were eligible.
Groups:
- Metformin + Insulin: 5 patients to continue on usual type 2 diabetic treatment consisting of 70/30 insulin, metformin and exercise and nutrition counseling.
  No Change
- Total: Total of all reporting groups
Arm/Group | Metformin + Insulin | QR-Bromocriptine +Metformin+Insulin | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (3) | 54 (3) | 50 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c
Description: Change from baseline HbA1c between subjects receiving QR-Bromocriptine + metformin + insulin compared to those subjects receiving metformin + insulin
Time Frame: Baseline - 24 weeks
Measure: Mean (Standard Error); unit: percent HbA1c
Groups:
- Metformin + Insulin: 5 patients to continue on usual type 2 diabetic treatment consisting of 70/30 insulin, metformin and exercise / nutrition counseling.
- QR-Bromocriptine + Metformin + Insulin: study drug add-on to usual therapy with insulin + metformin + exercise / nutritional counseling. The study drug is titrated up starting at one 0.8mg tab daily for 1 week, then 2 (0.8mg) tablets for week 2, then 3 tablets for week 3, then 4 tablets for week 4, then 5 tablets for week 5, then six tablets for week 6 (total 4.8). The titration was stopped when the patient reported side effects and the dose was subsequently reduced to the highest tolerable dose at which the side effect did not occur. The patient maintained this dose for the duration of the 24-week treatment period.
Arm/Group | Metformin + Insulin | QR-Bromocriptine + Metformin + Insulin
Number analyzed (Participants) | 5 | 7
percent HbA1c | 9.74 (0.56) | 7.98 (0.36)
Statistical Analysis 1: Comparison: Metformin + Insulin vs QR-Bromocriptine + Metformin + Insulin; Test type: Superiority or Other; p = 0.004, ANOVA

2. Secondary Outcome: Total Daily Insulin Dose
Description: Change in total daily insulin dose in patients treated with QR-Bromocriptine +metformin +insulin compared to metformin + insulin alone
Time Frame: Baseline - 24 weeks
Measure: Mean (Standard Error); unit: units of insulin
Arm/Group | Metformin + Insulin | QR-Bromocriptine + Metformin + Insulin
Number analyzed (Participants) | 5 | 7
units of insulin | 199 (33) | 147 (31)
Statistical Analysis 1: Comparison: Metformin + Insulin vs QR-Bromocriptine + Metformin + Insulin; Test type: Superiority or Other; p = 0.01, ANOVA
Statistical Analysis 2: Comparison: Metformin + Insulin vs QR-Bromocriptine + Metformin + Insulin; Test type: Superiority or Other; p = 0.009, ANOVA

ADVERSE EVENTS:
Arm/Group | Metformin + Insulin | QR-Bromocriptine + Metformin + Insulin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT01474018/Prot_SAP_000.pdf